CLINICAL TRIAL: NCT04043312
Title: A Randomized Controled Trial of Transcutaneous Magnetic Stimulation of the Stellate Ganglion to Treat Ventricular Tachycardia Storm
Brief Title: Magnetic Stimulation to Treat VT Storm
Acronym: STAR-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 833561
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Results first posted 2022-07-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Sham Comparator): Patients will receive one hour of sham stimulation.
  Interventions: Device: Magstim SuperRapid
- Active (Experimental): Patients will receive one hour of active magnetic stimulation to the left stellate ganglion.
  Interventions: Device: Magstim SuperRapid

INTERVENTIONS:
Device: Magstim SuperRapid — Transcutaneous magnetic stimulation targeting the left stellate ganglion.
  Arms: Active
Device: Magstim SuperRapid — Sham transcutaneous magnetic stimulation.
  Arms: Control

SUMMARY:
Ventricular Tachycardia storm is a medical emergency characterized by three or more episodes of ventricular arrhythmia within 24 hours and associated with a significantly increased mortality and massive health resource utilization. Several therapies are utilized including sympathetic blockade (through deep sedation and beta blockers), antiarrhythmic drugs, implantable cardioverter defibrillator (ICD) reprograming where applicable, and catheter ablation. Despite standard intervention, mortality rates remain high and additional therapeutic options are actively being investigated.

The overall objective of this proposal is to investigate whether transcutaneous magnetic stimulation designed to inhibit the left stellate ganglion can be used in this population. This is a single-center, randomized, sham-controlled trial to assess the efficacy of transcutaneous magnetic stimulation of the left stellate ganglion to treat patients with ventricular tachycardia storm.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3 episodes of VT in 24 hours

Exclusion Criteria:

* Pregnancy
* Implanted ventricular assist device
* Metal implanted in head or neck (except the mouth)
* Implanted medication pumps
* Cochlear implant
* Implanted brain stimulator
* Ocular implant
* History of active malignancy in region of stimulation (neck)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markman TM, Pothineni NVK, Zghaib T, Smietana J, McBride D, Amankwah NA, Linn KA, Kumareswaran R, Hyman M, Arkles J, Santangeli P, Schaller RD, Supple GE, Frankel DS, Deo R, Lin D, Riley MP, Epstein AE, Callans DJ, Marchlinski FE, Hamilton R, Nazarian S. Effect of Transcutaneous Magnetic Stimulation in Patients With Ventricular Tachycardia Storm: A Randomized Clinical Trial. JAMA Cardiol. 2022 Apr 1;7(4):445-449. doi: 10.1001/jamacardio.2021.6000. PMID 35171197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Active
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Active | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.6) | 66.9 (15.2) | 64.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26
Episodes of VT [Mean (Standard Deviation); unit: Episodes] | 14.8 (11.9) | 11.0 (8.7) | 12.7 (10.3)
Number of Antiarrhythmic Drugs Failed [Mean (Standard Deviation); unit: Drugs] | 2.2 (0.7) | 1.9 (0.5) | 2.0 (0.6)
Mechanical hemodynamic support [Count of Participants; unit: Participants] | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Ventricular Tachycardia - Incidence of Ventricular Tachycardia on Inpatient Telemetry Monitoring
Description: Incidence of ventricular tachycardia on inpatient telemetry monitoring
Time Frame: 24-hours following completion of the protocol
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 12 | 14
Participants | 7 | 4

2. Secondary Outcome: Cardioversion - Incidence of ICD Therapies or External Defibrillation Following Stimulation on Device Interrogation or Telemetry
Description: Incidence of ICD or external defibrillation following stimulation on device interrogation or telemetry
Time Frame: 48-hours following completion of the protocol
Population: Entire population
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 12 | 14
Participants | 7 | 4

3. Secondary Outcome: Number of Patients With Changes in ICD or Pacemaker Lead Impedances
Description: Number of patients with changes in lead impedance (unit: Ohms) on device interrogation
Time Frame: Immediately following completion of the protocol
Population: All patients with CIED
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

4. Secondary Outcome: Number of Patients With Changes in ICD or Pacemaker Lead Thresholds
Description: Number of patients with changes in lead thresholds (unit: mV) on device interrogation
Time Frame: Immediately following completion of the protocol
Population: Patients with CIED
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

5. Secondary Outcome: Number of Patient With Changes in ICD or Pacemaker Lead Sensitivities
Description: Number of patient with changes in lead sensitivity (unit: mA) on device interrogation
Time Frame: Immediately following completion of the protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

6. Secondary Outcome: Local Effect From Stimulation - Patient Reported Local Discomfort on Visual Analog Scale (0-10)
Description: Scores on a visual analog scale (0-10) of discomfort - 0= no discomfort, 1 = minimal discomfort, 10 = most severe discomfort imaginable.
Time Frame: Immediately following completion of the protocol
Population: Nonsedated patients
Measure: Mean (Standard Deviation); unit: Pain score
Arm/Group | Control | Active
Number analyzed (Participants) | 4 | 10
Pain score | 0 (0) | 0 (0)

7. Secondary Outcome: Antiarrhythmic Drugs Used Post Stimulation - Incidence of Antiarrhythmic Drug Use Post Stimulation Per Inpatient Medical Record
Description: Incidence of antiarrhythmic drug use post stimulation per inpatient medical record
Time Frame: 24 hours following completion of the protocol
Population: All participants
Measure: Mean (Standard Deviation); unit: Agents
Arm/Group | Control | Active
Number analyzed (Participants) | 12 | 14
Agents | 2.3 (0.8) | 0.9 (0.8)

8. Secondary Outcome: Number of Patients With Changes in ECG Parameters
Description: Number of patients with any clinical significant change in PR, QRS, or QT interval before and after stimulation.
Time Frame: Immediately following completion of the stimulation
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 12 | 14
Participants | 0 | 0

9. Secondary Outcome: Number of Patients With Changes in Vital Signs
Description: Number of patients with clinical significant change in heart rate or blood pressure during the procedure.
Time Frame: Immediately following the completion of the stimulation
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active
Number analyzed (Participants) | 12 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For 72 hours after enrollment
Arm/Group | Control | Active
All-Cause Mortality (participants affected / at risk) | 4/12 | 3/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT04043312/Prot_SAP_002.pdf